CLINICAL TRIAL: NCT00901212
Title: Evaluation fo Resynchronization Therapy for Heart Failure (EARTH)
Brief Title: Evaluation of Resynchronization Therapy for Heart Failure (EARTH)
Acronym: EARTH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Abbott Medical Devices (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Bernard Thibault, MD, Montreal Heart Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UCT-67914 (Greater Earth); 42560370
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; resynchronisation; ICD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LV Pacing (Active Comparator): left univentricular pacing
  Interventions: Device: Device programming
- BV Pacing (Active Comparator): biventricular pacing
  Interventions: Device: Device programming

INTERVENTIONS:
Device: Device programming — 6-month period

SUMMARY:
Heart failure is a major health problem in Canada. Recent advances in medical and device therapy have helped to reduce the morbidity and mortality of patients with this problem. Among these treatments, cardiac resynchronization therapy (CRT) has very recently been shown to be effective to improve functional class, quality of life and exercise tolerance of the patients with the most severe symptoms of heart failure and a prolonged duration of the QRS on the 12-lead Electrocardiography (ECG).

DETAILED DESCRIPTION:
Resynchronization of the failing ventricle is currently achieved by pacing the left and right ventricles simultaneously with specialized electrodes and a cardiac stimulator. However, controversy persists concerning the optimal configuration for cardiac pacing in these patients. Right ventricular pacing alone has been shown to be deleterious in some patient populations. The benefits of biventricular pacing in heart failure patients may be due primarily to left ventricular stimulation and may, in some patients, be decreased by the presence of simultaneous RV stimulation. Preliminary data from our own animal work suggest that in the majority of cases, LV stimulation alone is better than RV stimulation, and that BiV stimulation represents an intermediary situation between LV and RV stimulation.

ELIGIBILITY:
Inclusion Criteria (for Greater and Lesser EARTH):

Patient must answer "yes"

1. Does the patient require an ICD or an ICD replacement?
2. Does the patient have a documented LVEF less than or equal to 35% measured in the previous 6 months (without major concomitant clinical event)?
3. Does the patient have a QRS duration < 120 ms?
4. Is the patient in sinus rhythm?
5. Was the six-minute walk test distance less than 400 meters and limited by heart failure symptoms?

Exclusion Criteria:

Patient must have answered "NO" to all of the exclusion criteria

1. Does the patient have:

   * Indication for permanent ventricular pacing?
   * Chronotropic insufficiency?
   * Second or third degree AV block, either persistent or intermittent?
   * A pacemaker or an ICD which is paced in ventricular chamber more than 5% of the time?
2. Does the patient have a reversible cause of LV dysfunction such as post-partum cardiomyopathy, tachycardia induced cardiomyopathy, acute myocarditis or acute toxic cardiomyopathy (including acute alcoholic)?
3. Did the patient have myocardial infarction or cardiac surgery in the 6 weeks preceding the pre-implant visit?
4. Does the patient have a moderate or severe cardiac valve stenosis?
5. Is the patient's capacity to walk is limited by reasons other than heart failure symptoms (e.g., angina, intermittent claudication, severe lung condition or arthritis)?
6. Does the patient have severe coexisting illnesses making survival > 6 months unlikely?
7. Is the patient pregnant and/or nursing?
8. Is the patient unable or unwilling to consent or to comply with follow-up requirements?
9. Is the patient participating in another clinical study potentially interfering with the present trial?
10. Does the patient have a resynchronization system in place?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is total exercise duration at a constant submaximal load (ETT submaximal load is defined as 75% of peak exercise during the baseline metabolic evaluation) | one year

SECONDARY OUTCOMES:
Clinical, electrical, echocardiographic, MUGA scan endpoints, Neuro-hormones | one year

CONTACTS AND LOCATIONS:
Overall Officials: Bernard MD, Thibault, Study Chair — Montreal Heart Institute Research Center
Locations (11):
- Canada (11):
  - University of Alberta Hospital, Edmonton, Alberta
  - St-Paul's Hospital, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook & Women's Hospital, Toronto, Ontario
  - St-Michael's Hospital, Toronto, Ontario
  - CHUS-Fleurimont, Fleurimont, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM-Hôpital Hotel-Dieu, Montreal, Quebec
  - Sacre-Coeur Hospital, Montreal, Quebec
  - Institut Univ de Cardiologie et de Pneumologie de Québec, Québec, Quebec

REFERENCES:
- [Derived] Legris V, Thibault B, Dupuis J, White M, Asgar AW, Fortier A, Pitre C, Bouabdallaoui N, Henri C, O'Meara E, Ducharme A; EARTH Investigators. Right ventricular function and its coupling to pulmonary circulation predicts exercise tolerance in systolic heart failure. ESC Heart Fail. 2022 Feb;9(1):450-464. doi: 10.1002/ehf2.13726. Epub 2021 Dec 24. PMID 34953062
- [Derived] Thibault B, Ducharme A, Harel F, White M, O'Meara E, Guertin MC, Lavoie J, Frasure-Smith N, Dubuc M, Guerra P, Macle L, Rivard L, Roy D, Talajic M, Khairy P; Evaluation of Resynchronization Therapy for Heart Failure (GREATER-EARTH) Investigators. Left ventricular versus simultaneous biventricular pacing in patients with heart failure and a QRS complex >/=120 milliseconds. Circulation. 2011 Dec 20;124(25):2874-81. doi: 10.1161/CIRCULATIONAHA.111.032904. Epub 2011 Nov 21. PMID 22104549
- [Derived] Thibault B, Harel F, Ducharme A, White M, Frasure-Smith N, Roy D, Philippon F, Dorian P, Talajic M, Dubuc M, Gagne P, Guerra PG, Macle L, Rivard L, Khairy P. Evaluation of resynchronization therapy for heart failure in patients with a QRS duration greater than 120 ms (GREATER-EARTH) trial: rationale, design, and baseline characteristics. Can J Cardiol. 2011 Nov-Dec;27(6):779-86. doi: 10.1016/j.cjca.2011.03.010. Epub 2011 Jul 24. PMID 21791363